CLINICAL TRIAL: NCT03985397
Title: Evaluation of the Effect of Planned Discharge Training on Health Knowledge and Beliefs on Patients With Acute Myocardial Infarction
Brief Title: Patients With Acute Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Celal Bayar University (Other)
Responsible Party: Principal Investigator, Serap Tuna, internal medicine nursing lecturer doctor, Celal Bayar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20.478.486-332
Record Dates: First submitted 2019-05-27; First posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Cardiovascular Diseases
Keywords: discharge training; acute myocardial infarction; compliance to drug; compliance to diet; CARRF-KL.
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: The patients were randomly assigned to the intervention (50 patients) and control groups (50 patients) by lot according to the protocol numbers that are even and odd numbers (even numbers; the intervention group, odd numbers; the control group).
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (EG) (Experimental): At the first interview, after the application of the scales to the intervention group patients, planned discharge training and the manual prepared by the researcher were given. The second interview was performed 4 weeks later and the same scales were reapplied.
  Interventions: Other: discharge training
- Control group (No Intervention): In the first interview, scales were applied to the control group patients but planned discharge training was not given. The second interview was carried out 4 weeks later, and after the same scales were reapplied to the control group patients, planned discharge training was given. Therefore, the right of individuals to get education was not prevented.

INTERVENTIONS:
Other: discharge training — Providing planned discharge training according to the level of knowledge about diet, drug and individual monitoring compliance and cardiovascular risk factors of patients with acute myocardial infarction
  Arms: Experimental group (EG)

SUMMARY:
Aims and objectives The aim of this study was to determine whether planned discharge training given by the nurse has an impact on beliefs about cardiovascular disease risk factors knowledge level, compliance to drug therapy, compliance to diet and self- monitoring in patients with acute myocardial infarction (AMI).

Background: Increasing frequency of AMI, discharge of patients without discharge training cause recurrence of the disease and death.

Design: This study was done experimentally randomized controlled. Methods: The sample of the study includes 100 patients who were hospitalized due to AMI between September 2016 and December 2017 in coronary intensive care unit and cardiology department. The patients were divided into two groups according to random sampling method: intervention (n = 50) and control (n = 50) groups. Planned discharge training was given to the intervention group. Two interviews were conducted with each group with a one month break. The data of the research were collected by using the Patient Information Form, Beliefs about Medication Compliance Scale (BMCS), Beliefs about Dietary Compliance Scale (BDCS) and Beliefs about Self-Monitoring Scale (BSMS) and Cardiovascular Disease Risk Factors Knowledge Level (CARRF-KL) Scale.

DETAILED DESCRIPTION:
Cardiovascular diseases are one of the leading causes of mortality in all populations nowadays. Coronary artery disease (CAD) is considered to be the first cause of all deaths in the world. In 2017, 31% of the worldwide deaths (17.7 million) were caused by cardiovascular diseases. 80% of cardiovascular diseases are related to myocardial infarction (MI). It is thought that deaths due to cardiovascular diseases will reach 23.6 million in 2030.

Myocardial infarction is an irreversible heart muscle necrosis caused by prolonged ischemia. There are many factors that are effective in the formation of acute myocardial infarction (AMI). It is significant to know these factors that pose a risk to protection from this disease. Some of the risk factors can be changed and others include factors that are not possible to change. Risk factors that cannot be changed include individual features which are impossible to change; gender, age, family history, and presence of ACS in the history, biochemical or physiological features. In addition, risk factors that can be changed include obesity, low HDL-cholesterol level, high blood pressure, thrombogenic factors, hyperglycemia/diabetes mellitus, high plasma cholesterol, high plasma triglyceride level, stress, cholesterol-rich and high-calorie eating habits, smoking, consuming excess alcohol and sedentary life.

In patients with myocardial infarction, the mortality rate was 10% in the first years and 5% in the following years. Nurses play a significant role in the development, maintenance and prevention of diseases. Individuals with cardiovascular diseases should be given appropriate training before being discharged from the hospital. Training plan in patient/family education should be planned according to individual's readiness to learn, learning needs, education levels and previous experiences.

In the context of an effective training: in addition to basic information such as giving necessary information about the disease, cardiovascular risk factors and ways to reduce them, the importance of life change (drug use, healthy nourishment, smoking cessation, physical activity, etc.), regular policlinic control and guidance to cardiac rehabilitation program; information to meet the basic needs of the individual (return to work after MI, sexual life, housework, travel, driving, etc.) should be included. It is stated that the healing processes of the patients who are given discharge training have accelerated, and the number of recurrent applications to the hospital/policlinic has decreased and accordingly the patient care costs have decreased and the quality of care has increased.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction
* Discharge planned
* Minimal literacy
* 18-75 years of age
* No cancer or psychiatric diagnosis
* Not previously trained
* Being willing to participate in research

Exclusion Criteria:

* Patients who had myocardial infarction,
* İntubated, who had been intubated,
* were treated in other services due to additional diseases such as GIS bleeding, pneumonia, etc. after myocardial infarction,
* patients who had myocardial infarction and returned to their own services after treatment,
* who wanted to be transferred to another hospital while they were receiving treatment after myocardial infarction,
* who wanted to go to another hospital for an outpatient appointment,
* who did not want to come to polyclinic control from another city caused data loss.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Beliefs about Medication Compliance Scale | 5-10 minutes
  There are 12 sub-dimensions of the scale, namely benefit and disability; Items 1, 2, 7, 10, 11 measure the person's perception of benefit and items 3, 4, 5, 6, 8, 9, 12 measure the perception of obstacles. A higher score in the benefit subscale indicates that the perceived benefit is greater with behavior. The high score on the obstacles subscale shows that the subject perceives more of the obstacles when performing a behavior. The minimum total score of the scale is 12 and the maximum total score is 60.
Beliefs about Dietary Compliance Scale | 5-10 minutes
  It is a five-point Likert-type scale and consists of 12 items. There are two sub-dimensions: utility and obstacle. The first sub-dimension measures the individual's perception of benefit (items 1-5, 11, 12), and the second sub-dimension measures the perception of obstacles (items 6-10). The minimum total score of the scale is 12 and the maximum total score is 60.
Beliefs about Self-Monitoring Scale | 5-10 minutes
  Beliefs about Individual Follow-up Scale is a five-point Likert-type scale consisting of 18 items. There are two sub-dimensions: utility and obstacle. The benefits subscale (items 3, 5, 11, 15-17) showed that benefits were perceived more with higher scores; The high score in the obstacle subscale (items 1, 2, 4, 6-10, 12-14, 18) shows that the subject perceives more obstacles in conducting a behavior. The minimum total score of the scale is 18 and the maximum total score is 90.
Cardiovascular Disease Risk Factors Knowledge Level Scale. | 5-10 minutes
  The scale consists of 28 items. The first four of these items are the characteristics of cardiovascular diseases, 15 items are risk factors (5, 6, 9-12, 14, 18-20, 23-25, 27, 28 items), nine items (7, 8, 13, 15, 16, 17, 21, 22, 26) question the outcome of changes in risk behavior.
  The items in the scale are given as a complete sentence which can be true or false and they are asked to answer "Yes", "No" or iy I do not know ". Each correct answer is given 1 point. Twenty-two questions are scored straight and six questions (11, 12, 16, 17, 24, 26) are scored in the opposite direction. The highest total score that can be obtained from the scale is 28.

IPD SHARING:
Plan to Share IPD: No
I do not have a plan